CLINICAL TRIAL: NCT01883401
Title: Chronic Effects of Freeze-dried Strawberry Beverage on Cardiovascular Risk Factors in Subjects With Abdominal Adiposity and Dyslipidemia.
Brief Title: Chronic Effects of Freeze-Dried Strawberry Beverage on Cardiovascular Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University (Other)
Collaborators: University of Oklahoma (Other); California Strawberry Commission (Other)
Responsible Party: Principal Investigator, Arpita Basu, Assistant Professor, Oklahoma State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HE1015
Record Dates: First submitted 2013-05-13; First posted 2013-06-21 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Dyslipidemia; Obesity
Keywords: Strawberries; Heart health; Anthocyanins
MeSH Terms: conditions — Dyslipidemias; Obesity | interventions — Dietary Fiber

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- High dose strawberry (Experimental): 50g freeze-dried strawberries/day
  Interventions: Dietary Supplement: Freeze-dried strawberries
- Low-dose strawberry (Experimental): 25g freeze-dried strawberries/day
  Interventions: Dietary Supplement: Freeze-dried strawberries
- Fiber/calorie control (high dose) (Other): Dietary fiber (8g)
  Interventions: Dietary Supplement: Dietary fiber
- Fiber/calorie control (low dose) (Other): Dietary fiber (4g)
  Interventions: Dietary Supplement: Dietary fiber

INTERVENTIONS:
Dietary Supplement: Freeze-dried strawberries — 25g or 50g freeze-dried strawberries reconstituted in water
  Arms: High dose strawberry; Low-dose strawberry
Dietary Supplement: Dietary fiber — 4g or 8g dietary fiber blended in water
  Arms: Fiber/calorie control (high dose); Fiber/calorie control (low dose)

SUMMARY:
Berry anthocyanins have been shown to improve lipid profile in subjects with dyslipidemia while no such studies with whole strawberries have been reported in the US population. The investigators propose to examine the effects of low and high doses of freeze-dried strawberries on serum glucose, insulin, and lipid profile, biomarkers of oxidative stress and inflammation, in a 12-week randomized controlled trial. Subjects with abdominal adiposity and dyslipidemia (n=15/group) will be recruited at OUHSC and OSU, and randomly assigned to the low (25g/day) or high (50g/day) strawberry dose, or matched control (fiber and calories) group. The strawberry group will consume freeze-dried strawberry beverage (2 cups/day) and the controls will consume 2 cups beverage (fiber +calories) daily for 12 weeks. Blood draws, anthropometrics, blood pressure, and dietary data will be collected at screen, 6 and 12 weeks of the study to determine chronic and acute effects of strawberry intervention. Serum or plasma samples will be analyzed for fasting glucose, insulin, lipid profile including total cholesterol, LDL-, and HDL-cholesterol, triglycerides, lipid particle size, and levels of oxidative stress (malondialdehyde, oxidized LDL, myeloperoxidase), inflammation (high sensitivity C-reactive protein, adiponectin, interleukins) and adhesion molecules. Repeated measures ANOVA will be performed using a 5% significance level. We anticipate a dose response effect in decrease in lipids, oxidative stress or inflammation following strawberry intervention versus controls.

DETAILED DESCRIPTION:
The overall objective of this clinical trial is to investigate the effects of low and high doses of freeze-dried strawberries in cardiovascular risk factors in subjects with abdominal adiposity and dyslipidemia versus age and gender-matched controls.

ELIGIBILITY:
Inclusion Criteria:

* dyslipidemia
* abdominal adiposity (>35 inches for women, >40 inches for men)

Exclusion Criteria:

* on statin therapy
* taking hypoglycemic agents

Ages: 19 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Lipids (mg/dL) | 2.5 years
  Change in lipids and lipoproteins at screen and 12 weeks of the study

SECONDARY OUTCOMES:
Adhesion molecules (ng/mL) | 2.5 years
  Change in serum adhesion molecules (ICAM, VCAM) at screen and 12 weeks of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Arpita Basu, Phd, Principal Investigator — Oklahoma State University
Locations (1):
- Oklahoma State University, Stillwater, Oklahoma, United States

REFERENCES:
- [Background] Basu A, Fu DX, Wilkinson M, Simmons B, Wu M, Betts NM, Du M, Lyons TJ. Strawberries decrease atherosclerotic markers in subjects with metabolic syndrome. Nutr Res. 2010 Jul;30(7):462-9. doi: 10.1016/j.nutres.2010.06.016. PMID 20797478
- [Derived] Basu A, Betts NM, Nguyen A, Newman ED, Fu D, Lyons TJ. Freeze-dried strawberries lower serum cholesterol and lipid peroxidation in adults with abdominal adiposity and elevated serum lipids. J Nutr. 2014 Jun;144(6):830-7. doi: 10.3945/jn.113.188169. Epub 2014 Mar 26. PMID 24670970